CLINICAL TRIAL: NCT02404285
Title: A Multi-center, Double-blind, Vehicle-controlled Study to Evaluate the Clinical Effect of Daily Next Science™ Acne Gel (NAG) on Mild to Moderate Facial Acne
Brief Title: A Study to Evaluate the Clinical Effect of Daily Next Science™ Acne Gel (NAG) on Mild to Moderate Facial Acne
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Next Science TM (Industry)
Collaborators: Jacksonville Center For Clinical Research (Other); St. Johns Center for Clinical Research (Unknown); Fleming Island Center for Clinical Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSP-003
Record Dates: First submitted 2015-03-13; First posted 2015-03-31 (Estimated); Results first posted 2019-03-29 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vehicle (Placebo Comparator): Subjects will be treated with once daily vehicle and will attend screening, randomization, 2,4,8 and 12 week visits. The following will be assessed:
  1. Lesions will be counted and right, left and forward facing photographs will be taken
  2. Investigator Global Assessment
  3. Acne Quality of Life Questionnaire
  4. Treatment Area Assessment by Investigator
  Interventions: Drug: Vehicle
- NAG (Next Science Acne Gel) (Active Comparator): Subjects will be treated with once daily NAG and will attend screening, randomization, 2,4,8 and 12 week visits. The following will be assessed:
  1. Lesions will be counted and right, left and forward facing photographs will be taken
  2. Investigator Global Assessment
  3. Acne Quality of Life Questionnaire
  4. Treatment Area Assessment by Investigator
  Interventions: Drug: Next Science Acne Gel

INTERVENTIONS:
Drug: Next Science Acne Gel — Subjects will be instructed to apply a thin layer of the product to the entire face every evening after washing with Cetaphil cleanser and gently patting the skin dry. Product should not be applied around the eyes or near the mucous membranes. No other acne treatments will be applied to the face during study participation. Hands should be washed following application of study gel.
  Arms: NAG (Next Science Acne Gel)
Drug: Vehicle — Subjects will be instructed to apply a thin layer of the product to the entire face every evening after washing with Cetaphil cleanser and gently patting the skin dry. Product should not be applied around the eyes or near the mucous membranes. No other acne treatments will be applied to the face during study participation. Hands should be washed following application of study gel.
  Arms: Vehicle

SUMMARY:
This is a 12 week, multi-site, double-blind, vehicle-controlled study in subjects with mild to moderate facial acne. Subjects will be randomized 1:1 to apply either topical NAG or vehicle gel daily. Subjects will be evaluated for clinical acne and quality of life outcomes at baseline, 2 weeks, 4 weeks, 8 weeks and 12 weeks.

DETAILED DESCRIPTION:
Sample Size: N= 60 completed subjects Male and female subjects 12 years or older diagnosed with mild to moderate inflammatory facial acne vulgaris.

Subjects will be treated with once daily topical NAG or matching vehicle and will attend screening, randomization, 2,4,8 and 12 week visits. The following will be assessed:

1. Lesion counts with photography
2. Investigator Global Assessment
3. Acne Quality of Life Questionnaire
4. Treatment Area Assessment by Investigator

Subjects will discontinue all baseline topical acne treatments with a 2 week washout and/or all systemic acne treatments with a 3 week washout. All subjects will be provided open label Cetaphil facial cleanser and double-blind NAG or vehicle product.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ages 12 and above
2. Has 10 or more inflammatory lesions on the face (papules and pustules) as determined by qualified examiner at Start of Treatment.
3. In the area to be treated, has no significant facial dermatological conditions other than acne (as determined by the investigator) that would interfere with any study treatment or procedure
4. Is willing and able to discontinue use of all baseline acne treatments for the duration of their trial participation
5. Agrees to refrain from professional facial treatments during their trial participation.
6. Agrees to avoid tanning booth use and minimize sun exposure during their trial participation.
7. Is willing and able to follow instructions and procedures including attending scheduled study visits, which will require adequate transportation to the study site
8. Is able to read, understand and sign the informed consent document and communicate with study staff and investigator. If the subject is a minor, the parent or documented legal guardian must meet these consent requirements and the subject must be able to understand, agree to, and sign the assent form.

Exclusion Criteria:

1. Has more than 2 nodules/cystic acne lesions on the face
2. Has a history of significant reactions to topical acne treatments, or a known allergy or hypersensitivity to any listed ingredients
3. Has any history of skin malignancy
4. Has significant facial hair that would interfere with evaluation of acne lesions or global assessment.
5. Has used any systemic medications (including antibiotics, estrogens, retinoids) primarily for treatment of acne in the 21 days prior to randomization.
6. Has used estrogens primarily as treatment for acne in the 21 days prior to randomization (estrogens prescribed for other reasons will be allowed if stable for at least 30 days prior to randomization).
7. Has had any professional facial treatments in the 14 days prior to randomization.
8. Has received any investigational treatment in the 30 days prior to randomization.
9. Have any significant medical problems or other issues that would, in the investigator's judgment, affect their suitability for participation in this trial.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2015-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Greco, MD, Study Director — Jacksonville Center For Clinical Research; Annabelle Matias, MD, Principal Investigator — Fleming Island Center for Clinical Research; Lara Church, MD, Principal Investigator — St John's Center for Clinical Research
Locations (3):
- United States (3):
  - Fleming Island Center for Clinical Research, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - St. Johns Center for Clinical Research, Ponte Vedra, Florida

REFERENCES:
- [Result] Bernhardt MJ, Myntti MF. Topical Treatment With an Agent Disruptive to <em>P. acnes</em> Biofilm Provides Positive Therapeutic Response: Results of a Randomized Clinical Trial. J Drugs Dermatol. 2016 Jun 1;15(6):677-83. PMID 27272073

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were enrolled in the study after signing informed consent and meeting inclusion/exclusion criteria per protocol. A Washout period of 2-3 weeks was initiated for subjects discontinuing topical acne or systemic acne treatment respectively to normalize by washing their face twice a day with the study facial cleansing soap.
Groups:
- Vehicle: Subjects will be treated with once daily vehicle and will attend screening, randomization, 2,4,8 and 12 week visits. The following will be assessed:
  1. Lesions will be counted and right, left and forward facing photographs will be taken
  2. Investigator Global Assessment
  3. Acne Quality of Life Questionnaire
  4. Treatment Area Assessment by Investigator
  Vehicle: Subjects will be instructed to apply a thin layer of the product to the entire face every evening after washing with Cetaphil cleanser and gently patting the skin dry. Product should not be applied around the eyes or near the mucous membranes. No other acne treatments will be applied to the face during study participation. Hands should be washed following application of study gel.
- NAG (Next Science Acne Gel): Subjects will be treated with once daily NAG and will attend screening, randomization, 2,4,8 and 12 week visits. The following will be assessed:
  1. Lesions will be counted and right, left and forward facing photographs will be taken
  2. Investigator Global Assessment
  3. Acne Quality of Life Questionnaire
  4. Treatment Area Assessment by Investigator
  Next Science Acne Gel: Subjects will be instructed to apply a thin layer of the product to the entire face every evening after washing with Cetaphil cleanser and gently patting the skin dry. Product should not be applied around the eyes or near the mucous membranes. No other acne treatments will be applied to the face during study participation. Hands should be washed following application of study gel.
Period: Overall Study
Arm/Group | Vehicle | NAG (Next Science Acne Gel)
Started | 33 | 35
Completed | 31 | 33
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Vehicle: Subjects were treated with once daily vehicle and attended screening, randomization, 2,4,8 and 12 week visits. The following was assessed:
  1. Lesions were counted and right, left and forward facing photographs were taken
  2. Investigator Global Assessment
  3. Acne Quality of Life Questionnaire
  4. Treatment Area Assessment by Investigator
  Vehicle: Subjects were instructed to apply a thin layer of the product to the entire face every evening after washing with Cetaphil cleanser and gently patting the skin dry. Product should was not to be applied around the eyes or near the mucous membranes. No other acne treatments was applied to the face during study participation.
- NAG (Next Science Acne Gel): Subjects were treated with once daily vehicle and attended screening, randomization, 2,4,8 and 12 week visits. The following was assessed:
  1. Lesions were counted and right, left and forward facing photographs were taken
  2. Investigator Global Assessment
  3. Acne Quality of Life Questionnaire
  4. Treatment Area Assessment by Investigator
  Next Science Acne Gel: Subjects were instructed to apply a thin layer of the product to the entire face every evening after washing with Cetaphil cleanser and gently patting the skin dry. Product should was not to be applied around the eyes or near the mucous membranes. No other acne treatments was applied to the face during study participation.
- Total: Total of all reporting groups
Arm/Group | Vehicle | NAG (Next Science Acne Gel) | Total
Number analyzed (Participants) | 33 | 35 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 35 | 68
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 40
  Male | 14 | 14 | 28
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33 | 35 | 68

OUTCOME MEASURES:

1. Primary Outcome: Change in Inflammatory Lesions With Daily Use of NAG Compared With Vehicle After 12-weeks of Use.
Description: Percent change in number of Inflammatory lesions with daily use of NAG compared with vehicle after 12-weeks of use.
Time Frame: Baseline until 12 weeks
Population: Subjects who completes all visits.
Measure: Mean (Standard Error); unit: % change of inflammatory lesions count
Groups:
- Vehicle: Subjects were treated with once daily vehicle and the following was assessed at baseline, 2,4,8 and 12 week visits:
  1. Lesions were counted and right, left and forward facing photographs were taken
- NAG (Next Science Acne Gel): Subjects were treated with once daily NAG and the following was assessed at baseline, 2,4,8 and 12 week visits:
  1. Lesions were counted and right, left and forward facing photographs were taken
Arm/Group | Vehicle | NAG (Next Science Acne Gel)
Number analyzed (Participants) | 33 | 35
% change of inflammatory lesions count | -27 (12.5) | -44 (8.6)
Statistical Analysis 1: Comparison: Vehicle vs NAG (Next Science Acne Gel); Test type: Superiority; p < 0.01, ANOVA

2. Secondary Outcome: Percent Change in Non-Inflammatory Lesion Counts After 12 Weeks of Treatment.
Description: Percent Change in Number of Non-inflammatory lesions (open and closed comedones) were counted after 12 weeks of either Vehicle of NAG treatment
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: % Change Non-inflammatory lesion count
Groups:
- Vehicle: Subjects will be treated with once daily vehicle and the following were assessed at baseline, 2,4,8 and 12 week visits:
  1. Lesions will be counted and right, left and forward facing photographs will be taken
  2. Investigator Global Assessment
  3. Acne Quality of Life Questionnaire
  4. Treatment Area Assessment by Investigator
  Vehicle: Subjects will be instructed to apply a thin layer of the product to the entire face every evening after washing with Cetaphil cleanser and gently patting the skin dry. Product should not be applied around the eyes or near the mucous membranes. No other acne treatments will be applied to the face during study participation. Hands should be washed following application of study gel.
- NAG (Next Science Acne Gel): Subjects will be treated with once daily NAG and and the following was assessed at baseline, 2,4,8 and 12 week visits:
  1. Lesions will be counted and right, left and forward facing photographs will be taken
  2. Investigator Global Assessment
  3. Acne Quality of Life Questionnaire
  4. Treatment Area Assessment by Investigator
  Next Science Acne Gel: Subjects will be instructed to apply a thin layer of the product to the entire face every evening after washing with Cetaphil cleanser and gently patting the skin dry. Product should not be applied around the eyes or near the mucous membranes. No other acne treatments will be applied to the face during study participation. Hands should be washed following application of study gel.
Arm/Group | Vehicle | NAG (Next Science Acne Gel)
Number analyzed (Participants) | 33 | 35
% Change Non-inflammatory lesion count | -6.5 (7.1) | -34.1 (5.8)

3. Secondary Outcome: Final Investigator Global Assessment Score With Daily Use of NAG Compared With Vehicle After 12-weeks.
Description: Change in Investigator Global Assessment (IGA) score (0-5) with daily use of NAG compared with vehicle after 12-weeks. IGA score is worse at 5, with improvement at lower scores (best at 0).
Time Frame: Baseline until 12 weeks
Measure: Mean (Standard Error); unit: Score on a scale
Groups:
- Vehicle: Subjects were treated with once daily vehicle and attended baseline, 2,4,8 and 12 week visits and the number of non-inflammatory lesions were counted.
- NAG (Next Science Acne Gel): Subjects were treated with once daily NAG and attended baseline, 2,4,8 and 12 week visits and the number of non-inflammatory lesions were counted.
Arm/Group | Vehicle | NAG (Next Science Acne Gel)
Number analyzed (Participants) | 33 | 35
Score on a scale
  Mean at Baseline | 2.8 (.08) | 2.4 (.09)
  Mean after 12 Weeks | 2.3 (0.13) | 2.0 (0.14)
Statistical Analysis 1: Comparison: Vehicle vs NAG (Next Science Acne Gel); Test type: Superiority; p < 0.001, ANOVA

4. Secondary Outcome: Change in Erythema Scores With Daily Use of NAG Compared With Vehicle After 12-weeks.
Description: Change in Erythema (measure of redness) scores with daily use of NAG compared with vehicle after 12-weeks.Treatment area evaluation scoring system ranges from 0-3, with 0 being Absent (none) and 3 being Severe (intense, marked presence).
Time Frame: Baseline until 12 weeks
Population: The Next Science Acne Gel had average erythema score decreasing from 0.5 to 0.3 for the Acne Gel and to 0.5 to 0.4 for the Vehicle Control (not shown).
Measure: Mean (Standard Deviation); unit: Average Score on a scale
Arm/Group | Vehicle | NAG (Next Science Acne Gel)
Number analyzed (Participants) | 33 | 35
Average Score on a scale
  Mean at Baseline | .5 (.8) | .5 (.7)
  Mean after 12 weeks | 0.4 (0.8) | 0.3 (0.5)

5. Secondary Outcome: Change in Dryness With Daily Use of NAG Compared With Vehicle After 12-weeks.
Description: Change in Dryness score with daily use of NAG compared with vehicle after 12-weeks. Treatment area evaluation scoring system ranges from 0-3, with 0 being Absent (none) and 3 being Severe (intense, marked presence).
Time Frame: Baseline until 12 weeks
Population: NAG application yielded Dryness average scores decreasing from 0.3 to 0.1 over 12 weeks compared to no decrease in the Vehicle control (0.3 to 0.3).
Measure: Mean (Standard Deviation); unit: Average score on a scale
Groups:
- Vehicle: Subjects will be treated with once daily vehicle and will attend baseline, 2,4,8 and 12 week visits. The following will be assessed:
  1. Lesions will be counted and right, left and forward facing photographs will be taken
  2. Investigator Global Assessment
  3. Acne Quality of Life Questionnaire
  4. Treatment Area Assessment by Investigator
  Vehicle: Subjects will be instructed to apply a thin layer of the product to the entire face every evening after washing with Cetaphil cleanser and gently patting the skin dry. Product should not be applied around the eyes or near the mucous membranes. No other acne treatments will be applied to the face during study participation. Hands should be washed following application of study gel.
- NAG (Next Science Acne Gel): Subjects will be treated with once daily NAG and will attend baseline, 2,4,8 and 12 week visits. The following will be assessed:
  1. Lesions will be counted and right, left and forward facing photographs will be taken
  2. Investigator Global Assessment
  3. Acne Quality of Life Questionnaire
  4. Treatment Area Assessment by Investigator
  Next Science Acne Gel: Subjects will be instructed to apply a thin layer of the product to the entire face every evening after washing with Cetaphil cleanser and gently patting the skin dry. Product should not be applied around the eyes or near the mucous membranes. No other acne treatments will be applied to the face during study participation. Hands should be washed following application of study gel.
Arm/Group | Vehicle | NAG (Next Science Acne Gel)
Number analyzed (Participants) | 33 | 35
Average score on a scale
  Mean at Baseline | .3 (.5) | .3 (.5)
  Mean after 12 Weeks | 0.3 (0.5) | 0.1 (0.5)

6. Secondary Outcome: Change in Burning/Stinging With Daily Use of NAG Compared With Vehicle After 12-weeks.
Description: Change in Burning/Stinging scores with daily use of NAG compared with vehicle after 12-weeks. Treatment area evaluation scoring system ranges from 0-3, with 0 being Absent (none) and 3 being Severe (intense, marked presence).
Time Frame: Baseline until 12 weeks
Population: NAG application resulted in average Burning or Stinging scores increasing from 0.0 to 0.1 over 12 weeks, compared to a decrease in Vehicle Control from 0.1 to 0.0.
Measure: Mean (Standard Deviation); unit: Average score on a scale
Arm/Group | Vehicle | NAG (Next Science Acne Gel)
Number analyzed (Participants) | 33 | 35
Average score on a scale
  Mean at Baseline | .1 (.3) | 0 (0)
  Mean after 12 Weeks | 0 (0.3) | 0.1 (0.3)

7. Secondary Outcome: Change in Erosion With Daily Use of NAG Compared With Vehicle After 12-weeks.
Description: Change in Erosion scores with daily use of NAG compared with vehicle after 12-weeks. Treatment area evaluation scoring system ranges from 0-3, with 0 being Absent (none) and 3 being Severe (intense, marked presence).
Time Frame: Baseline until 12 weeks
Population: NAG application resulted in average scores remaining between 0.1 and 0.0 for all time points for both NAG and Vehicle groups.
Measure: Mean (Standard Deviation); unit: Average score on a scale
Arm/Group | Vehicle | NAG (Next Science Acne Gel)
Number analyzed (Participants) | 33 | 35
Average score on a scale
  Mean at Baseline | 0 (0) | 0 (0)
  Mean after 12 Weeks | 0 (0.1) | 0 (0.1)

8. Secondary Outcome: Change in Edema With Daily Use of NAG Compared With Vehicle After 12-weeks.
Description: Change in Edema scores with daily use of NAG compared with vehicle after 12-weeks. Treatment area evaluation scoring system ranges from 0-3, with 0 being Absent (none) and 3 being Severe (intense, marked presence).
Time Frame: Baseline until 12 weeks
Population: NAG application resulted in average scores decreasing from 0.1 to 0.0 for the Acne Gel, and from 0.2 to 0.1 for the Vehicle Control.
Measure: Mean (Standard Deviation); unit: Average score on a scale
Arm/Group | Vehicle | NAG (Next Science Acne Gel)
Number analyzed (Participants) | 33 | 35
Average score on a scale
  Mean at Baseline | .2 (.4) | 0.1 (.3)
  Mean after 12 Weeks | 0.1 (0.4) | 0 (0.3)

9. Secondary Outcome: Change in Pain With Daily Use of NAG Compared With Vehicle After 12-weeks.
Description: Change in Pain scores with daily use of NAG compared with vehicle after 12-weeks. Treatment area evaluation scoring system ranges from 0-3, with 0 being Absent (none) and 3 being Severe (intense, marked presence).
Time Frame: Baseline until 12 weeks
Population: NAG and vehicle application yielded average pain scores decreasing from 0.1 to 0.0.
Measure: Mean (Standard Deviation); unit: Average score on a scale
Arm/Group | Vehicle | NAG (Next Science Acne Gel)
Number analyzed (Participants) | 33 | 35
Average score on a scale
  Mean at Baseline | .1 (.2) | .1 (.4)
  Mean at 12 Weeks | 0 (0.3) | 0 (0.3)

10. Secondary Outcome: Change in Itching With Daily Use of NAG Compared With Vehicle After 12-weeks.
Description: Change in Itching scores with daily use of NAG compared with vehicle after 12-weeks. Treatment area evaluation scoring system ranges from 0-3, with 0 being Absent (none) and 3 being Severe (intense, marked presence).
Time Frame: Baseline until 12 weeks
Population: NAG application resulted in Itching scores of 0.1 to 0.0 for the Acne Gel and from 0.2 to 0.0 for the Vehicle Control.
Measure: Mean (Standard Deviation); unit: Average score on a scale
Arm/Group | Vehicle | NAG (Next Science Acne Gel)
Number analyzed (Participants) | 33 | 35
Average score on a scale
  Mean at Baseline | .2 (.5) | .1 (.3)
  Mean at 12 Weeks | 0 (0.3) | 0 (0.3)

11. Other Pre Specified Outcome: Change in Quality of Life - Self Perception With Daily Use of NAG Compared With Vehicle After 12-weeks.
Description: Change in Self Perception scores with daily use of NAG compared with vehicle after 12-weeks. The Acne Quality of Life (QoL) Questionnaire Form was used to determine the practical improvements in quality of life. The Acne-QoL form is a validated measure that contains 19 questions referring to the past week, organized into four area: self-perception, role-social, role-emotional, and acne symptoms. Each question gauges how much acne affects the subject, with answers ranging from 0 (extremely) to 6 (not at all). Domain scores are calculated by taking the average scores within each domain, with high scores reflecting better QoL determination. The number of subjects with a negative score for each quality of life region was determined at each time-point. Those with a negative score, were those with a score of 3.5 or less, indicating that the disease was having a meaningful effect on their lives.
Time Frame: Baseline until 12 weeks
Population: The average self-perception score for NAG users increased from 4.1 to 5.0.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Vehicle | NAG (Next Science Acne Gel)
Number analyzed (Participants) | 33 | 35
Score on a scale
  Mean at Baseline | 3.5 (2.1) | 4.1 (1.9)
  Mean at 12 Weeks | 4.6 (1.5) | 5.0 (1.5)

12. Other Pre Specified Outcome: Change in Quality of Life - Role Emotional With Daily Use of NAG Compared With Vehicle After 12-weeks.
Description: Change in Role-Emotional scores with daily use of NAG compared with vehicle after 12-weeks. At baseline and each subsequent visit, subjects completed the Acne-QoL form after being given verbal instructions by the study coordinator. The Acne QoL is a validated measure that contains 19 questions referring to the past week, organized into four areas: self-perception, role-social, role-emotional, and acne symptoms. Each question gauges how much acne affects the subject, with answers ranging from 0 (extremely) to 6 (not at all). Domain scores are calculated by taking the average scores within each domain, with high scores reflecting better QoL determination. The number of subjects with a negative score for each quality of life region was determined at each time-point. Those with a negative score, were those with a score of 3.5 or less, indicating that the disease was having a meaningful effect on their lives
Time Frame: Baseline until 12 weeks
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Vehicle | NAG (Next Science Acne Gel)
Number analyzed (Participants) | 33 | 35
Score on a scale
  Mean at Baseline | 3.9 (1.6) | 3.9 (1.8)
  Mean at 12 Weeks | 4.6 (1.4) | 4.8 (1.3)

13. Other Pre Specified Outcome: Change in Quality of Life - Perceived Acne Symptoms With Daily Use of NAG Compared With Vehicle After 12-weeks.
Description: Change in the subjects perception of their acne symptoms with daily use of NAG compared with vehicle after 12-weeks. At baseline and each subsequent visit, subjects completed the Acne-QoL form after being given verbal instructions by the study coordinator. The Acne QoL is a validated measure that contains 19 questions referring to the past week, organized into four areas: self-perception, role-social, role-emotional, and acne symptoms. Each question gauges how much acne affects the subject, with answers ranging from 0 (extremely) to 6 (not at all). Domain scores are calculated by taking the average scores within each domain, with high scores reflecting better QoL determination. The number of subjects with a negative score for each quality of life region was determined at each time-point. Those with a negative score, were those with a score of 3.5 or less, indicating that the disease was having a meaningful effect on their lives
Time Frame: Baseline until 12 weeks
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Vehicle | NAG (Next Science Acne Gel)
Number analyzed (Participants) | 33 | 35
Score on a scale
  Mean at Baseline | 3.4 (1.1) | 3.4 (1.2)
  Mean at 12 Weeks | 4.4 (1.3) | 4.5 (1.1)

14. Other Pre Specified Outcome: Change in Quality of Life - Role Social With Daily Use of NAG Compared With Vehicle After 12-weeks.
Description: Change in subjects social response to their acne with daily use of NAG compared with vehicle after 12-weeks. At baseline and each subsequent visit, subjects completed the Acne-QoL form after being given verbal instructions by the study coordinator. The Acne QoL is a validated measure that contains 19 questions referring to the past week, organized into four areas: self-perception, role-social, role-emotional, and acne symptoms. Each question gauges how much acne affects the subject, with answers ranging from 0 (extremely) to 6 (not at all). Domain scores are calculated by taking the average scores within each domain, with high scores reflecting better QoL determination. The number of subjects with a negative score for each quality of life region was determined at each time-point. Those with a negative score, were those with a score of 3.5 or less, indicating that the disease was having a meaningful effect on their lives
Time Frame: Baseline until 12 weeks
Population: The average Role-Social score increased from 4.5 to 5.3.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Vehicle | NAG (Next Science Acne Gel)
Number analyzed (Participants) | 33 | 35
Score on a scale
  Mean at Baseline | 4.1 (2.0) | 4.5 (2.0)
  Mean at 12 Weeks | 4.7 (1.7) | 5.3 (1.6)

ADVERSE EVENTS:
Time Frame: 12 Weeks.
Groups:
- Vehicle: Subjects were treated with once daily vehicle and attended screening, randomization, 2,4,8 and 12 week visits. The following was assessed:
  1. Lesions were counted and right, left and forward facing photographs were taken
  2. Investigator Global Assessment
  3. Acne Quality of Life Questionnaire
  4. Treatment Area Assessment by Investigator
  Vehicle: Subjects were instructed to apply a thin layer of the product to the entire face every evening after washing with Cetaphil cleanser and gently patting the skin dry.
- NAG (Next Science Acne Gel): Subjects were treated with once daily NAG and attended screening, randomization, 2,4,8 and 12 week visits. The following was assessed:
  1. Lesions were counted and right, left and forward facing photographs were taken
  2. Investigator Global Assessment
  3. Acne Quality of Life Questionnaire
  4. Treatment Area Assessment by Investigator
  Next Science Acne Gel: Subjects were instructed to apply a thin layer of the product to the entire face every evening after washing with Cetaphil cleanser and gently patting the skin dry.
Arm/Group | Vehicle | NAG (Next Science Acne Gel)
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/35
Other Adverse Events (participants affected / at risk) | 7/33 | 9/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle (N=33) | NAG (Next Science Acne Gel) (N=35)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Gastritis (General disorders) | 1 (1) | 0 (0)
Vomiting (General disorders) | 1 (1) | 0 (0) — Vomiting
Haemtoma (Infections and infestations) | 1 (1) | 0 (0) — Left Thumbnail Haematoma
Rhinitis (Infections and infestations) | 2 (2) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 1 (1)
General aches (General disorders) | 0 (0) | 1 (1)
Mild celiac disease (General disorders) | 0 (0) | 1 (1)
Abdominal cramps (General disorders) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Cough (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 1 (1)
Otitis Media (Infections and infestations) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No